CLINICAL TRIAL: NCT05004441
Title: Fruquintinib Combined With mFOLFOX6/FOLFIRI in First-line Treatment for Metastatic Colorectal Cancer：HCCSC C02 Trial
Brief Title: Fruquintinib Combined With mFOLFOX6/FOLFIRI in First-line Treatment for Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Fuxiang (Other)
Collaborators: Hubei Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Xiangya Hospital of Central South University (Other); Huangshi Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhou Fuxiang, Professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC C02
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line treatment (Experimental): First-line treatment: Fruquintinib Combined With mFOLFOX6/FOLFIRI for twelve cycles.
  Maintenance treatment: Fruquintinib and Capecitabine
  Interventions: Drug: Fruquintinib Combined With mFOLFOX6/FOLFIRI

INTERVENTIONS:
Drug: Fruquintinib Combined With mFOLFOX6/FOLFIRI — Fruquintinib (3mg) will be given p.o. daily

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Fruquintinib Combined With mFOLFOX6/FOLFIRI as the first-line treatment of Metastatic Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ≤75 years
2. Histologically confirmed unresectable or metastatic stage colorectal cancer
3. Known RAS activating mutation/wild type and BRAF wild type;
4. Patients have not received systematic treatment for unresectable or metastatic colorectal cancer (those who have received adjuvant or neoadjuvant chemotherapy with one regimen and relapsed more than 12 months after the end of chemotherapy can be enrolled);
5. At least one measurable disease according to RECIST 1.1 guidelines for solid tumors；
6. BMI≥18；
7. ECOG 0-1
8. Life expectancy > 12 weeks
9. Patients must have adequate organ function
10. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration;
11. Informed consent has been signed.

Exclusion Criteria:

1. Have received other systemic anti-tumor therapies within 2 weeks before recruited(eg.chemotherapy or radiotherapy, immunotherapy, biological or hormonal therapy, or any VEGFR inhibitor treatment);
2. Known BRAF activating mutation
3. systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs; Or patients need more than two antihypertensive drugs;
4. Clinically significant electrolyte abnormality;
5. Proteinuria ≥ 2+ (1.0g/24hr);
6. Patients have untreated central nervous system metastasis;
7. Patients have not recovered from all toxicities associated with prior anti-tumor therapy ,to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE v5.0) Grade of 0 or 1, except for alopecia and oxaliplatin induced neurotoxicity ≤ 2 , and the previous surgery did not recover completely;
8. Have received other systemic anti-tumor therapies within 4 weeks before recruited;
9. Clinical uncontrolled active infections, such as acute pneumonia and active hepatitis B / C (previous history of hepatitis B virus infection, whether drug controlled or not, HBV DNA ≥ 104) × Copy number or ≥ 2000 IU / ml);
10. Dysphagia or known malabsorption of drugs;
11. Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI;
12. Have evidence or history of bleeding tendency within 2 months after enrollment, the researcher assessed that moderate or severe bleeding tendency was not suitable for enrollment;
13. Stroke (including transient ischemic attack) occurred within 12 months before admission;
14. Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
15. Pregnant or lactating women;
16. Allergic to fruquintinib；
17. History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation;
18. Patients with acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before admission; Or a history of arterial thrombosis or deep venous thrombosis;
19. There are concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger the safety of patients or affect the completion of the study, or any laboratory abnormalities that are not suitable for participating in the clinical trial according to the judgment of the researcher,
20. Serious psychological or mental disorders that may affect the compliance study;
21. Participating in other drug clinical trials within 4 weeks before recruited.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 36 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
disease control rate (DCR) | 36 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Progression-Free Survival (PFS) | 36 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
overall survival (OS) | 36 months
  OS is the time from enrollment to death due to any cause.
adverse events (AE) | 36 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No